CLINICAL TRIAL: NCT02871999
Title: Clinical Trial on Acupuncture Adjuvant Treatment in the Pain After the Surgery of Gastrointestinal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaonan Cui (Other)
Responsible Party: Sponsor-Investigator, Xiaonan Cui, Professor, Chief Physician, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCKY2016-39
Record Dates: First submitted 2016-08-03; First posted 2016-08-18 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Gastrointestinal Carcinoma; Pain
Keywords: Acupuncture Therapy; Pain degree after surgery
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): This group receives normal treatment after surgery,with no acupuncture.
  Interventions: Procedure: Laparoscopic Surgery
- Experimental group (Experimental): This group receives acupuncture therapy besides normal treatment after surgery. The acupuncture therapy starts after 24 hours of surgery, 1 time a day, 30 minutes every time, until the fifth day.
  Interventions: Device: Acupuncture therapy; Procedure: Laparoscopic Surgery

INTERVENTIONS:
Device: Acupuncture therapy
  Arms: Experimental group
Procedure: Laparoscopic Surgery

SUMMARY:
Clinical trial on acupuncture adjuvant treatment in the pain after the surgery of gastrointestinal carcinoma. Gastrointestinal cancer patients are diagnosed by pathology or cell biology. Patients are randomized into 2 groups: The control group receive normal treatment only, the experimental group receive acupuncture therapy besides normal treatment. Clinical evaluation is based on the observation of the pain degree and life quality improvement. Blood biochemistry tests mainly include Prostaglandin E2(PGE2),5-hydroxytryptamine(5-HT), histamine(HIS), malondialdehyde (MDA), superoxide dismutase (SOD), glutathione peroxidase (GSH-Px), adrenaline, nor-adrenaline, tumor necrosis factor (TNF)-α, cell flow cytometry on Th1, Th2, Th17, Treg cytokines as well as serum cortisol, estradiol (female), progesterone (female), testosterone (male) etc.

ELIGIBILITY:
Inclusion Criteria:

1. General anesthesia,Gastric and Colorectal Cancer surgery under Laparoscopic;
2. Pathology diagnosed;
3. Brain, heart, lung, liver, kidney are at good condition before surgery;
4. No mental disorder, no conscious obstacle, no limbs disability.

Exclusion Criteria:

1. Severely complication after surgery;
2. Contraindication of the acupuncture;
3. Patients with mental disease;
4. Patients taking part in other clinical trials, being treated with other biotherapy or immunotherapy and researchers consider not suitable for clinical subjects for other reasons will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Pain degree change after surgery, Graded according to Numerical Rating Scale(NRS) | day 1, day 2, day 3, day 4, day 5, day 6, day 7 after surgery

SECONDARY OUTCOMES:
Assessing the quality of life(QOL) change in 4 grades and recording: appetite, mental state, sleep, fatigue, attitude towards treatment, daily life ability | day 1, day 2, day 3, day 4, day 5, day 6, day 7 after surgery
Prostaglandin E2(PGE2) in blood | day 2,day 7 after surgery
Estradiol(Female) in blood | day 2, day 7 after surgery
Th1/Th2 in blood | day 2, day 7 after surgery
5-Hydroxytryptamine(5-HT) in blood | day 2,day 7 after surgery
Histamine(HIS) in blood | day 2,day 7 after surgery
Th17/Treg in blood | day 2, day 7 after surgery
Testosterone(Male) in blood | day 2,day 7 after surgery

IPD SHARING:
Plan to Share IPD: Undecided